CLINICAL TRIAL: NCT06716918
Title: The Effect of Antenatal Corticosteroids Prior to Planned Cesarean Section in Early Term on Neonatal Hypoglycemia
Brief Title: Effect of Antenatal Corticosteroids on Neonatal Hypoglycemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Bahgat Heshmat, Resident doctor, Assiut University
Other Study IDs: Antenatal corticosteroids
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Antenatal Corticosteroids
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients took antenatal corticosteroids prior to planned cesarean section
  Interventions: Drug: Corticosteroid Injection
- patients didnt't take antenatal corticosteroids prior to planned cesarean section

INTERVENTIONS:
Drug: Corticosteroid Injection — Participants who have received antenatal corticosteroids (betamethasone or dexamethasone) prior to cesarean section as part of their prenatal care.
  Groups: patients took antenatal corticosteroids prior to planned cesarean section

SUMMARY:
Comparing the incidence of neonatal hypoglycemia in infants born to mothers who received antenatal corticosteroids to those who did not.

DETAILED DESCRIPTION:
Antenatal corticosteroids (ACS) are widely used to enhance fetal lung maturation in pregnancies at risk of preterm birth. However, their role in early-term pregnancies (37 to 38 weeks gestation) prior to planned cesarean section has been gaining attention. Early-term neonates delivered by cesarean section are at an increased risk of respiratory complications, and studies have shown that ACS can reduce these risks by accelerating fetal lung development. The use of ACS in this population, however, has raised concerns about its potential effects on neonatal metabolic outcomes, particularly neonatal hypoglycemia.

Neonatal hypoglycemia, a common metabolic disorder in the early postnatal period, is often associated with antenatal corticosteroid exposure. ACS may increase fetal insulin production by stimulating pancreatic beta cells, leading to an increased risk of hypoglycemia after birth. Research indicates that while ACS effectively reduces respiratory morbidity in early-term neonates, it may concurrently raise the risk of neonatal hypoglycemia. For instance, a meta-analysis found a significant association between ACS and an increased incidence of hypoglycemia in term and near-term infants.

Given these findings, research is crucial to assess the balance of risks and benefits of ACS in early-term cesarean deliveries. While ACS appears to reduce respiratory complications, understanding its full impact on neonatal hypoglycemia will help guide its use in clinical practice

ELIGIBILITY:
Inclusion Criteria:

- 1. Women with singleton pregnancies at 37-38 weeks of gestation (early-term) scheduled for planned cesarean sections.

2. Participants who have received antenatal corticosteroids prior to cesarean section as part of their prenatal care.

Exclusion Criteria:

* 1. Women delivering before 37 weeks or after 39 weeks of gestation would be excluded, as the study focuses on early-term deliveries.

  2. Women with any form of diabetes, including pre-existing type 1 or type 2 diabetes, and gestational diabetes. This ensures that the study focuses on non-diabetic populations, as diabetes can independently affect neonatal glucose regulation and complicate the assessment of hypoglycemia risk due to corticosteroids.

  3. Women with severe maternal health such as preeclampsia, chronic hypertension, or other systemic illnesses, might be excluded to avoid confounding variables.

  4. Women who did not complete the full course of antenatal corticosteroids may be excluded, as the effect of partial doses could differ from complete treatment.

  5. Women with multiple gestations (e.g., twins or triplets) may be excluded due to the added complexity of multiple-birth pregnancies and their unique risk.

  6. Neonates with known congenital anomalies, genetic disorders, or other pre-existing medical conditions that could affect glucose metabolism

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women Health Hospital, Faculty of medicine, Assiut university
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Comparing the incidence of neonatal hypoglycemia in infants born to mothers who received antenatal corticosteroids to those who did not.. | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital, Faculty of medicine, Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Melamed N, Asztalos E, Willan AR, et al. Neonatal hypoglycemia following administration of antenatal corticosteroids: A systematic review and meta-analysis. J Obstet Gynaecol Can. 2017;39(1):36-45.
- [Background] Stutchfield PR, Whitaker R, Gliddon AE, Hobson L, Kotecha S, Doull IJ. Behavioural, educational and respiratory outcomes of antenatal betamethasone for term caesarean section (ASTECS trial). Arch Dis Child Fetal Neonatal Ed. 2013 May;98(3):F195-200. doi: 10.1136/archdischild-2012-303157. Epub 2013 Feb 19. PMID 23424017
- [Background] Kamath-Rayne BD, Rozance PJ, Goldenberg RL, Jobe AH. Antenatal corticosteroids beyond 34 weeks gestation: What do we do now? Am J Obstet Gynecol. 2016 Oct;215(4):423-30. doi: 10.1016/j.ajog.2016.06.023. Epub 2016 Jun 21. PMID 27342043
- [Background] Magro-Malosso ER, Saccone G, Di Tommaso M, Mele M, Berghella V. Neuraxial analgesia to increase the success rate of external cephalic version: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2016 Sep;215(3):276-86. doi: 10.1016/j.ajog.2016.04.036. Epub 2016 Apr 27. PMID 27131581